CLINICAL TRIAL: NCT00228228
Title: T-Cell Vaccination in the Treatment of Probable Multiple Sclerosis
Brief Title: TCV -01-002: T-Cell Vaccination in the Treatment of Probable Multiple Sclerosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-01-2490-AA-CTIL
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2006-08-29 (Estimated); Status verified 2006-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; T-cell vaccination; Autoreactive T cells
MeSH Terms: conditions — Multiple Sclerosis

INTERVENTIONS:
Biological: T cell vaccination

SUMMARY:
In the present study, we, the investigators at Sheba Medical Center, intend to evaluate T cell vaccination (TCV) in patients with probable multiple sclerosis (MS) within up to 3 months after the first clinical attack. It is of the utmost importance to evaluate the treatment effects at the onset of disease, i.e. in patients with probable MS, in order to evaluate whether early treatment can prevent the second attack (conversion to definite MS). Moreover, at disease onset, the immunological process of epitope spreading associated with the exposure of the immune system to myelin antigens is still limited. With additional attacks, increased recognition of new self-determinants of encephalitogenic peptides presented to the immune system during the inflammatory process occurs, and enhances further disease activity. The aim of the early TCV treatment approach is to stop this process as early as possible, during the onset of the disease, thus preventing additional attacks and disease progression.

We will evaluate the effect of TCV on clinical, immunological and magnetic resonance imaging (MRI) parameters in patients with probable MS.

DETAILED DESCRIPTION:
Inclusion criteria:

* Age: 15 - 50 years.
* Three months within the acute onset of neurological symptoms suggestive of the first attack of multiple sclerosis.
* Diagnosis of CPMS C3 (Poser criteria).
* Positive brain MRI according to Fazekas criteria.
* Negative pregnancy test and use of effective contraceptive for female patients who are sexually active.
* Signed written informed consent.

Exclusion criteria:

* Blood tests suggestive of other autoimmune diseases.
* Known allergic reactions to MRI contrast media.
* A clear regression of the neurological symptoms after the first attack that suggests a primary-progressive course.
* Corticosteroid treatment in the previous 4 weeks (28 days).
* Previous treatment with immunosuppressive medications such as cyclophosphamide, azathioprine, methotrexate, mitoxantrone or cyclosporine.
* Previous treatment with interferon beta 1a or 1b, copolymer-1, IVIg, plasmapheresis.

ELIGIBILITY:
Inclusion Criteria:

* Ages 15-50
* Three months within the acute onset of neurological symptoms suggestive of multiple sclerosis
* Diagnosis of clinically probable MS (CPMS) C3: 1 attack with at least 1 clinical manifestation in addition to positive brain MRI as defined in the protocol, signifying paraclinical evidence (Poser criteria 1983).
* Positive Brain MRI: at least 4 focal lesions involving the white matter of 3 lesions if one is periventricular > 3mm diameter, each
* Negative pregnancy test and use of effective contraceptives for female patients who are sexually active.
* Signed written informed consent.

Exclusion Criteria:

* Blood tests suggestive of other autoimmune diseases
* Known allergic reaction to MRI contrast media.
* A clear regression of the neurological symptoms after the first attack that excludes a primary progressive course.
* Corticosteroid treatment in the previous 4 weeks.
* Previous treatment with immunosuppressive medications such as cyclophosphamide, azathioprine, methotrexate, mitoxantrone, or cyclosporine.
* Previous treatment with interferon beta 1a or 1b copolymer-1 IVIg, plasmapheresis.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80
Dates: Start 2002-05; Study Completion 2006-12

PRIMARY OUTCOMES:
The rate of progression to definite MS (second attack) during the study
Time to progression to definite MS (second attack)

SECONDARY OUTCOMES:
Change in the count of new gadolinium (GD) enhancing lesions from two baseline (B) MRIs to the final (F) MRIs
Change in total volume of new GD enhancing lesions from two baseline MRIs (B) to the final MRIs (F)
The change in neurological disability as measured by the Expanded Disability Status Scale (EDSS)

CONTACTS AND LOCATIONS:
Overall Officials: Anat Achiron, MD, PhD, Principal Investigator — Multiple Sclerosis Center, Sheba Medical Center, Tel-Hashomer, Israel; Mathilda Mandel, MD, Principal Investigator — Blood Bank, Sheba Medical Center, Tel-Hashomer, Israel
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel